CLINICAL TRIAL: NCT00808964
Title: Phase 2 Study of NU172 Anticoagulation in Patients Undergoing Coronary Artery Bypass Graft Surgery OFF-Pump
Brief Title: Study of NU172 as Anticoagulation in Patients Undergoing Off-pump CABG Surgery
Acronym: SNAP-CABG-OFF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: ARCA Biopharma, Inc. (Industry)
Responsible Party: Michael Bristow, M.D., PhD, ARCA biopharma, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: CLINPRO-303
Record Dates: First submitted 2008-12-12; First posted 2008-12-16 (Estimated); Last update posted 2011-06-10 (Estimated); Status verified 2011-06

CONDITIONS: Heart Disease
Keywords: CABG; anticoagulant; Off-Pump CABG
MeSH Terms: conditions — Heart Diseases | interventions — NU172

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: NU172 — NU172 administered IV bolus followed by continuous infusion during CABG surgery

SUMMARY:
This is a Phase 2, multicenter, open-label, single-arm, sequential cohort study to be conducted in up to 30 subjects. The study will evaluate subjects undergoing primary, elective, off-pump CABG surgery with median sternotomy.

ELIGIBILITY:
Inclusion Criteria:

* Must give written informed consent prior to initiation of any study related procedures
* Male or female subjects at least 18 years of age
* Subject is accepted for primary, elective off-pump CABG surgery with planned sternotomy without other planned concomitant cardiac surgical procedures
* New York Heart Association (NYHA) Class III or less heart failure
* Available for follow-up assessments

Exclusion Criteria:

* Prior surgery with median sternotomy
* Prior CABG surgery
* Women of childbearing potential who are not using adequate contraceptive precautions (e.g. intrauterine device, oral contraceptives,barrier methods, or other contraception deemed adequate by the investigator); women who are pregnant or lactating
* Stroke within the previous 6 months
* History of stroke with residual neurological deficit
* Intracranial neoplasm, arteriovenous malformation or aneurysm
* Any prior exposure to NU172
* Contraindication to unfractionated heparin
* Refusal to undergo blood transfusion, should it be necessary
* Symptomatic gout
* Serum uric acid >11mg/dL at screening
* Known bleeding diathesis
* Known thrombotic diathesis
* Participation in any study of an investigational device, drug or biologic within 30 days prior to planned surgery
* Any other disease or condition that, in the judgment of the investigator would interfere with the subject's ability to comply with study procedures and requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Safety and efficacy of NU172 in patients undergoing off-pump CABG surgery | 30 day follow-up visit

SECONDARY OUTCOMES:
Evaluate the pharmacokinetic (PK)profile of NU172 in patients undergoing off-pump CABG surgery | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Smedira, M.D., Principal Investigator — The Cleveland Clinic